CLINICAL TRIAL: NCT00552799
Title: Randomised Controlled Trial to Investigate Whether Prophylactic Antibiotics Can Prevent Further Episodes of Cellulitis (Erysipelas) of the Leg (PATCH I)
Brief Title: RCT to Investigate if Prophylactic Antibiotics Prevent Further Episodes of Cellulitis (Erysipelas) of the Leg
Acronym: PATCH1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Action Medical Research (Other); UK Dermatology Clinical Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06002; ISRCTN34716921; EudraCT No. 2006-000381-36
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Cellulitis/Erysipelas of the Leg
Keywords: cellulitis; lymphoedema; penicillin; clinical trial
MeSH Terms: conditions — Cellulitis; Lymphedema | interventions — Penicillin V

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Penicillin VK 250 mg b.d.
  Interventions: Drug: Penicillin VK
- 2 (Placebo Comparator): placebo tablet b.d.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Penicillin VK — Biconcave tablet 250mg oral, b.d.
  Arms: 1
Other: placebo — biconcave tablet matching active comparator as much as possible in size and shape
  Arms: 2

SUMMARY:
To assess whether a period of prophylactic penicillin after an episode of cellulitis of the leg reduces the risk of repeat episodes. Participants are randomised to receive 12 months of prophylaxis (penicillin VK 250mg b.d. or placebo). The PATCH I study will recruit only patients with recurrent disease.

DETAILED DESCRIPTION:
Cellulitis of the leg is an common, acute, painful and potentially serious infection of the skin and subcutaneous tissue. It currently accounts for 2-3% of UK hospital admissions. The average length of in-patient stay is 9 days (Hospital Episode Statistics, Department of Health (UK), 2002-2003) and 25-50% of treated patients suffer further episodes and other morbidity, such as oedema and ulceration.

Cellulitis of the lower leg is usually due to streptococcal infection that has entered into the body via a relatively subtle portal, such as toeweb fissures. Penicillin is the most useful of the commonly used oral antibiotics against streptococci, although other agents such as flucloxacillin are often used if staphylococcal infection is a clinical possibility.

There are numerous risk factors for cellulitis of the lower leg and recurrent disease is one the biggest problems.

Existing evidence for the use of prophylactic antibiotics to prevent further episodes is very limited. Two small randomised controlled trials (RCTs) hint at possible benefit, but these studies are very small (16 and 40 participants respectively). Despite this, many physicians routinely use prophylactic antibiotics for recurrent cellulitis, although opinions on the value of such practice is firmly divided.

This study will recruit over a 12-24 month period participants who have completed the therapy for the current episode of cellulitis. Participants will be followed up for up to 24 months with telephone calls at 10 days, 3 months, 6 months, 9 months and 12 months and then every 6 months after completing the intervention. A diary will also be provided as an "aid memoir" to phone calls and to note missed tablets and recurrence of cellulitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cellulitis of either leg AND a history of at least one previous episode of cellulitis of either leg within the three

Exclusion Criteria:

Any doubt about the certainty of the diagnosis of either the index episode or the previous episode (if applicable), will be grounds for exclusion. Additionally, patients with any of the following will be excluded:

* Taken antibiotic prophylaxis (defined as more than 3 months usage) for the prevention of cellulitis within 6 months prior to index episode.
* A time lapse of longer than 12 weeks since the start of treatment for the index episode to the date of potential randomisation into the trial.
* Known allergy to penicillin.
* Preceding leg ulceration, surgery or penetrating trauma, as these cases are more likely to be caused by staphylococcal infection. (NB: this does not exclude patients with toeweb maceration/tinea pedis or other minor/blunt wounds).
* Treating physician or principal investigator unwilling to randomise patient. This includes, but is not limited to:

  * The treating physician and/or patient feels that prophylactic antibiotics are not in the patient's best interests and therefore entry to this study would be inappropriate.
  * The treating physician and/or patient feels it would not be ethical or appropriate for the patient to receive placebo and so they are not willing/able to accept randomisation
  * Concomitant medication that would mean that long-term penicillin is inappropriate
  * Diagnostic uncertainty
  * Gastrointestinal disease causing persistent diarrhoea or vomiting severe enough to affect the absorption of the phenoxymethylpenicillin.
  * Allergic diathesis or severe bronchial asthma severe enough to preclude the use of phenoxymethylpenicillin.
  * Confounding concurrent disease (e.g. DVT).
* No access to a telephone.
* Aged less than 16 years.
* Unable to give informed consent.
* Already taking part in a research study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2006-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is time to next episode of cellulitis | variable

SECONDARY OUTCOMES:
Secondary outcomes include: i) the proportion of participants with repeat episodes of cellulitis; ii) proportion of participants with oedema and/or ulceration; iii) cost-effectiveness; iv) predictors of response (multiple regression model). | variable

CONTACTS AND LOCATIONS:
Overall Officials: Hywel Williams, Professor, Study Director — University of Nottingham
Locations (25):
- South Infirmary-Victoria University Hospital, Cork, Ireland
- United Kingdom (24):
  - Queens Medical Centre, Nottingham, Nottinghamshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Amersham Hospital, Amersham
  - Brighton General Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - Cumberland Infirmary, Carlisle
  - Derbyshire Royal Infirmary, Derby
  - University Hospital of North Durham, Durham
  - Gloucestershire Royal Infirmary, Gloucester
  - James Paget University Hospital, Great Yarmouth
  - Princess Royal Hospital, Hull
  - Ipswich Hospital, Ipswich
  - Queen Elizabeth Hospital, Kings Lynn
  - Leicester Royal Infirmary, Leicester
  - Broadgreen Hospital, Liverpool
  - Altnagelvin Area Hospital, Londonderry
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Royal Berkshire Hospital, Reading
  - Hope Hospital, Salford
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Watford General Hospital, Watford
  - York Hospital, York